CLINICAL TRIAL: NCT02766244
Title: Indocyanine Green (ICG) and SPY Imaging for Assessment of Burn Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Principal Investigator, Sharmila Dissanaike, Professor, Texas Tech University Health Sciences Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 003 NCT02028520; NCT02028520 (obsolete NCT alias)
Record Dates: First submitted 2015-11-13; First posted 2016-05-09 (Estimated); Results first posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ICG/SPY (Experimental): Daily wound care with antibiotic ointments after cleansing plus evaluation using ICG/SPY fluorescence.
  Interventions: Device: ICG/SPY; Drug: Antibiotic Ointment

INTERVENTIONS:
Device: ICG/SPY — indocyanine green fluorescence imaging
Drug: Antibiotic Ointment — Antibiotic ointment

SUMMARY:
Three patients were recruited for assessment of ICG fluorescence in burns.

DETAILED DESCRIPTION:
The early determination of healing potential in indeterminate thickness burns may be difficult to establish by visual inspection alone, even for experienced burn practitioners. This case series explores the use of indocyanine green (ICG) fluorescence using portable bedside assessment as a potential tool for early determination of burn depth. Three subjects with indeterminate thickness burns had daily perfusion assessment using ICG fluorescence assessment using the SPY machine (SPY®, Lifecell Corp., NJ, USA) in addition to standard burn care. The fluorescence was quantified as a percentage of the perfusion of intact skin, and areas of hypo and hyper-perfusion were indicated. The burn surgeon, blinded to the ICG results, made a clinical determination of the need for skin grafting or discharge. The perfusion in areas of differing depth of burn were compared over the entire study period to determine both the magnitude of difference, and the point in the time course of healing when these changes became evident.

ELIGIBILITY:
Inclusion Criteria:

* patients with burn less than 15% TBSA

Exclusion Criteria:

* none

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dissanaike S, Abdul-Hamed S, Griswold JA. Variations in burn perfusion over time as measured by portable ICG fluorescence: A case series. Burns Trauma. 2014 Oct 25;2(4):201-5. doi: 10.4103/2321-3868.142397. eCollection 2014. PMID 27602383

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ICG/SPY
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ICG/SPY
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Size of burn [Median (Full Range); unit: % of body surface area] | 7 [7 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Perfusion of Burned Area
Description: Perfusion as measured by ICG Fluorescence
Time Frame: 5 days
Measure: Number; unit: % perfusion compared to normal skin
Groups:
- Patient 1 Superficial; Patient 1 Deep Tissue; Patient 2 Superficial; Patient 2 Deep Tissue; Patient 3 Superficial; Patient 3 Deep Tissue: Daily wound care with antibiotic ointments after cleansing plus evaluation using ICG/SPY fluorescence.
  ICG/SPY: indocyanine green fluorescence imaging
  Antibiotic Ointment: Antibiotic ointment
Arm/Group | Patient 1 Superficial | Patient 1 Deep Tissue | Patient 2 Superficial | Patient 2 Deep Tissue | Patient 3 Superficial | Patient 3 Deep Tissue
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
% perfusion compared to normal skin
  Day 1 | 200 | 100 | 205 | 180 | 205 | 110
  Day 2 | 300 | 200 | 210 | 110 | 180 | 190
  Day 3 | 250 | 180 | 280 | 200 | 500 | 380
  Day 4 | 180 | 100 | 470 | 250 | 200 | 150
  Day 5 | 205 | 140 | NA — No data on this day | NA — No data on this day | NA — No data on this day | NA — No data on this day

ADVERSE EVENTS:
Time Frame: Three months
Arm/Group | ICG/SPY
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No